CLINICAL TRIAL: NCT04232449
Title: Oral Corticosteroids for Post-infectious Cough in Adults: A Double-blind Randomised Placebo-controlled Trial in Swiss Family Practices (OSPIC Trial)
Brief Title: Oral Corticosteroids for Post-infectious Cough in Adults
Acronym: OSPIC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: too few patients were included
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-02214; ex16Zeller
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Post-infectious Cough
Keywords: Upper Respiratory Tract Infection; oral corticosteroid treatment; Cough-related Quality of Life (QoL)
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: multi-centre, 1:1 randomised, parallel-group, placebo-controlled, superiority trial with blinded patients, physicians and outcome assessors in a primary health care setting
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: blinded patients, physicians and outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Identically looking, numbered and marked medication glass jars with 5 daily doses of 40 mg (2 tablets of 20 mg) of prednisone (intervention group) are provided by General Physicians (GPs) to participants. PREDNISON Galepharm Tabl. 20 mg are manufactured according to Good Manufacturing Practice (GMP)-guidelines.
  The prednisone medication is manufactured by Galepharm AG, 8700 Küsnacht (ZH) and packaged and labelled by the Hospital Pharmacy of the University Hospital Basel. The PREDNISON tablets' active substance is Prednisonum; the tablets also contain Excipiens pro compresso. Swissmedic authorization 50821
  Interventions: Drug: PREDNISON Galepharm Tabl. 20 mg
- Control group (Placebo Comparator): Identically looking, numbered and marked medication glass jars with 5 daily doses of placebo (control group) are provided by General Physicians (GPs) to participants.
  The content of the placebo tablets is as follows: Lactose monohydrate 140 mg, microcrystalline cellulose 68 mg, Croscarmellose sodium 5 mg, Magnesium stearate 2mg. The placebo tablets were manufactured by Apotheke Hotz, Zürichstrasse 176, CH- 8700 Küsnacht.
  Interventions: Drug: placebo tablets

INTERVENTIONS:
Drug: PREDNISON Galepharm Tabl. 20 mg — 5 daily- doses of 40 mg (2 tablets of 20 mg) of prednisone
  Arms: Intervention group
Drug: placebo tablets — 5 daily- doses of placebo (2 tablets)
  Arms: Control group

SUMMARY:
The purpose of this study is to assess whether a 5-day treatment with orally administered prednisone provides patient-relevant benefits by improving the cough-related QoL of patients with post-infectious cough triggered by an Upper Respiratory Tract Infection (URTI) and seeking care in adult primary care practices. The study aims to describe an efficacy and safety profile for a 5-day prednisone treatment compared to a 5-day course of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeing a GP for a dry or productive post-infectious cough (3 to 8 weeks) after Upper Respiratory Tract Infection (URTI)
* Patients able and willing to give informed consent by themselves and to fill in the LCQ on day 0 with the GP and to answer phone calls from the research staff/study nurse at day 7, 14, and 28, and at 3 months for outcome assessment

Exclusion Criteria:

* Patients with known or suspected diagnoses associated with cough, such as: pneumonia or suggestive symptoms and signs (abnormal vital signs, i.e. heart rate >100/min, respiratory rate >25/min, fever), allergic rhinitis, sinusitis, bronchial asthma, chronic pulmonary disease (COPD), or gastroesophageal reflux disease,
* Patients with other chronic disease such as bronchiectasis, cystic fibrosis, cancer, tuberculosis, heart failure.
* Use of inhaled or oral corticosteroids within the last four weeks
* Immunodeficiency/immunocompromised state (e.g. cancer chemotherapy, HIV infection, administration of immune-suppressive agents)
* Pregnancy/ breastfeeding
* Regular treatment known to be associated with cough (e.g. angiotensin converting enzyme inhibitors)
* Patients with pharmacotherapy for glaucoma or osteoporosis
* Experienced fractures due to osteoporosis
* Patients with uncontrolled diabetes (as deemed by GPs who appraise whether the potential side effects of short-time corticosteroids on glucose levels exceed the hypothesised benefit on cough)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Cough-related Quality of Life (QoL) assessed by the Leicester Cough Questionnaire (LCQ) score | assessment done 14 days after randomisation
  The LCQ comprises 19 items and takes 5 to 10 minutes to complete. The LCQ is a validated QoL measurement tool for non-specific cough and assesses the impact of cough on various aspects of life, including emotions, sleeping behaviour, work and relationships. It contains 19 items which are divided over 3 domains: physical (8 items), psychological (7 items) and social (4 items), with a 7-point Likert response scale.

SECONDARY OUTCOMES:
Change in Cough-related QoL assessed by the LCQ score | assessment done at 7 and 28 days and at 3 months after randomisation
  The LCQ comprises 19 items and takes 5 to 10 minutes to complete. The LCQ is a validated QoL measurement tool for non-specific cough and assesses the impact of cough on various aspects of life, including emotions, sleeping behaviour, work and relationships. It contains 19 items which are divided over 3 domains: physical (8 items), psychological (7 items) and social (4 items), with a 7-point Likert response scale.
Overall cessation of cough | assessment done 7, 14, 28 days and 3 months after randomization
  Overall cessation of cough (yes/ no)
Incidence rate of re-consultations with the treating GP and/or hospitalisations | within 3 months following randomisation
  Incidence rate of re-consultations with the treating General Physician (GP) and/or hospitalisations
Total Adverse Events (number) | within 3 months after randomization
  Total Adverse Events (number)
Serious Adverse Events (number) | within 3 months after randomization
  Serious Adverse Events (number)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Zeller, Prof. Dr. med, Principal Investigator — Centre for Primary Health Care (uniham-bb); University of Basel
Locations (2):
- Switzerland (2):
  - Centre for Primary Health Care (uniham-bb); University of Basel; Kantonsspital Baselland, Liestal
  - Institute of Primary and Community Care, University of Lucerne, Lucerne

REFERENCES:
- [Derived] Merlo C, Essig S, Brancati-Badarau DO, Leuppi JD, Speich B, Erlanger TE, Hemkens LG, Zeller A. Oral corticosteroids for post-infectious cough in adults: study protocol for a double-blind randomized placebo-controlled trial in Swiss family practices (OSPIC trial). Trials. 2020 Nov 23;21(1):949. doi: 10.1186/s13063-020-04848-4. PMID 33225983